CLINICAL TRIAL: NCT01703897
Title: Evaluation of Esophageal Pressures and Reflux in Obese Patients Before and During Anesthesia Using High-resolution Solid-state Manometry
Brief Title: Esophageal Manometry and Impedance Study in Obese Patients Before and During Anesthesia
Status: Withdrawn | Type: Observational
Sponsor: Örebro University, Sweden (Other)
Responsible Party: Principal Investigator, Alex de Leon, MD, PhD, Örebro University, Sweden
Other Study IDs: Linde-Imped
Record Dates: First submitted 2012-10-08; First posted 2012-10-11 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Obesity
Keywords: gastric by-pass surgery
MeSH Terms: conditions — Obesity | interventions — Manometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Obese patients
  Interventions: Device: Manometry and Impedance analysis

INTERVENTIONS:
Device: Manometry and Impedance analysis

SUMMARY:
The purpose of this study is to evaluate the effects of anesthesia on the esophageal body in obese patients before and during anesthesia.

DETAILED DESCRIPTION:
Obesity is an increasing heath problem in western countries and is associated with increased risks during anesthesia.

Using high-resolution solid-state manometry the investigators aim to study esophageal pressures and measure the incidence of regurgitation of gastric contents during anesthesia induction in obese patients. The investigators aim to include 16 obese patients, with BMI > 35, undergoing laparoscopic gastric by-pass.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients
* aged 18-60 years
* BMI>35
* ASA classification I-III

Exclusion Criteria:

* Use of drugs that interfere with esophageal motility
* Gastro-esophageal reflux disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Obese patients
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-10

PRIMARY OUTCOMES:
Esophageal pressures after laparoscopic gastric by pass | 2 years after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Intensive care, University Hospital of Örebro, Örebro, Sweden